CLINICAL TRIAL: NCT00176696
Title: Detection of Nociception ("Pain") During General Anesthesia
Brief Title: Biobehavioral Recovery From Surgery and Anesthesia
Status: Terminated | Type: Observational
Why Stopped: Principal Investigator has left the UMDNJ
Sponsor: University of Medicine and Dentistry of New Jersey (Other)
Responsible Party: Sponsor
Organization: Rutgers, The State University of New Jersey (Other)
Other Study IDs: 0120050013
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2016-10-06 (Estimated); Status verified 2008-06

CONDITIONS: Pain, Postoperative
Keywords: general anesthesia; pain; depth of anesthesia
MeSH Terms: conditions — Pain, Postoperative; Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Use of FACE monitor and BIS monitor — Face monitor records facial muscle activity
  Other Names: BIS (Bispectral Score)determines the depth of anesthesia

SUMMARY:
Reducing postoperative pain leads to increased patient comfort and facilitates speedy recovery and discharge from the hospital following surgery. The focus of controlling postoperative pain has gradually shifted from postoperative management to intraoperative management. The investigators believe that this study is a unique opportunity to assess the adequacy of intraoperative analgesia, allowing for immediate administration of the appropriate opioid analgesics. The purpose of this research is to bring to light the applicability of facial electromyography as an intraoperative solution to postoperative pain management.

DETAILED DESCRIPTION:
After consenting to enter the study, the subject will be asked a series of questions regarding his/her medical history. He/she will be shown the test for determining consciousness by squeezing the experimenter's hand when asked. It will be explained to him/her that once unconscious, he/she will not be able to respond to the command of squeezing the hand. The facial monitor will be shown to the patient, as well as its location of placement.

Intraoperative Period: The leads will be placed for the FACE monitor as well as for the BIS monitoring device. The objective of the BIS monitor which is already in use in the University Hospital Operating room suites is to determine consciousness. An identical and typical anesthetic protocol will be utilized for all the patients in order to eliminate anesthetic factors. The protocol is as follows:

After administration of propofol for induction, a forearm tourniquet device will be inflated to a pressure greater than 200 mm Hg. A muscle relaxant will then be given once the tourniquet is inflated while the arm with the tourniquet will not be paralyzed. This allows for a check on the unconsciousness of the patient; that is, the patient will be told, "squeeze my hand". It is expected that no patient will respond by squeezing his or her hand because they are unconscious and anesthetized. The maximum length of time the cuff will be inflated is 20 minutes. Tourniquets applied to the entire leg or arm are normally inflated for up to 120 minutes and are standard practice in orthopedic surgery.

One group of patients, determined randomly, will be administered 250 ug of fentanyl during induction of anesthesia, while the second group, also determined randomly, will be administered 50 ug of fentanyl. Both groups of patients will be administered an inhalational anesthetic (isoflurane, desflurane, or sevoflurane) at the level 30% above that which insures unconsciousness (called 1.1 MAC), but will not be given nitrous oxide during the 10 minutes of our study period due to this gas' effect on Hagihira's "loss of bicoherence" phenomenon.

The study period will begin 5 minutes before surgical incision, and will end 5 minutes after surgical incision. Our hypothesis is that central registration of pain exists despite the presence of adequate unconsciousness in the patient, and FACE technology will complement the use of the BIS (EEG) monitor to ensure effective administration of anesthesia for patients in the future.

ELIGIBILITY:
Inclusion Criteria:

* Subjects 18-65 years of age
* Subjects who are English speaking
* Subjects undergoing surgery in the supine position
* Subjects who are undergoing a procedure where the surgical incision is expected to be at least 4 inches
* Subjects who are undergoing a surgical procedure below the level of their arms.
* Female subjects who have a negative Sure-Vue pregnancy test.
* Subjects who are undergoing surgery under general anesthesia.

Exclusion Criteria:

* If the scheduled surgery involves the head, neck or arms.
* Subjects who have a history of chronic pain
* Subjects who have cognitive disabilities secondary to medical, chemical and genetic causes.
* Subjects who have peripheral vascular disease of the arms.
* Subjects who have carpal tunnel syndrome.
* Subjects who have psychiatric, substance abuse and cognitive impairments
* Subjects who have had a stroke which has affected function of the upper extremities
* Subjects who have had a mastectomy or other type of surgery which may have affected the lymph nodes of the arms
* Subjects who do not have a telephone
* Subjects who are having surgery under nerve block or regional anesthesia
* Subjects who are pregnant
* Subjects who have an electrical source, i.e. pacemaker or defibrillator

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: subjects undergoing surgery
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2005-08; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
detection of pain during general anesthesia | after induction of anesthesia

SECONDARY OUTCOMES:
Visual analogue scale for first two days post anesthesia | 2 post op days

CONTACTS AND LOCATIONS:
Overall Officials: Henry L. Bennett, PhD, Principal Investigator — Rutgers, The State University of New Jersey

IPD SHARING:
Plan to Share IPD: No